CLINICAL TRIAL: NCT03898895
Title: Combination of Radiotherapy With Anti-PD-1 Antibody for Unresectable Biliary Tract Cancer
Acronym: CORRECT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming Kuang, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTC002
Record Dates: First submitted 2019-03-30; First posted 2019-04-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Biliary Tract Cancer; Radiotherapy; Immunotherapy
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiotherapy+anti-PD-1 antibody (Experimental): The total radiation dose is over 45Gy without damaging organic function. Conventional intensity-modulated radiotherapy or stereotactic body radiation therapy are both allowed. Camrelizumab 200mg intravenously every 3 weeks will be initiated within 7 days after radiotherapy. Patients will receive camrelizumab until clinical or radiographic disease progression, unacceptable toxicity, death or withdrawal. If disease progression is confirmed by radiologic examinations, another 200mg camrelizumab should be applied to the patient, then another radiologic examination will be performed 4 weeks later to confirm or exclude progression. If progression is confirmed, the camrelizumab should be stopped.
  Interventions: Combination Product: Radiotherapy+anti-PD-1 antibody

INTERVENTIONS:
Combination Product: Radiotherapy+anti-PD-1 antibody — The total radiation dose is over 45Gy without damaging organic fucntion. Conventional intensity-modulated radiotherapy or stereotactic body radiation therapy are both allowed. Camrelizumab 200mg intravenously every 3 weeks will be initiated within 7 days after radiotherapy. Patients will receive camrelizumab until clinical or radiographic disease progression, unacceptable toxicity, death or withdrawal. If disease progression is confirmed by radiologic examinations, another 200mg camrelizumab should be applied to the patient, then another radiologic examination will be performed 4 weeks later to confirm or exclude progression. If progression is confirmed, the camrelizumab should be stopped.
  Other Names: RT/IO

SUMMARY:
The study is a single-arm, phase II trial. The purpose is to investigate both the efficacy and safety of radiotherapy combined with anti-PD-1 antibody in unresectable biliary tract cancer patients.

DETAILED DESCRIPTION:
The trial will recruit 36 patients, and they will undergo radiotherapy plus anti-PD-1 antibody. Patients will receive conventional intensity-modulated radiotherapy or stereotactic body radiation therapy first for a total dose more than 45Gy. Camrelizumab 200mg intravenously every 3 weeks will be initiated within 7 days after radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 75 years old;
2. Histopathologically confirmed unresectable primary or initial postoperative recurrent BTC without distant metastasis;
3. No previous radiotherapy or systemic therapy;
4. Adequate volume of the uninvolved liver (larger than 700 mL);
5. At least one measurable lesion based on Response Evaluation Criteria in Solid Tumors 1.1 criteria;
6. Eastern Cooperative Oncology Group performance status score of 0 or 1;
7. Adequate hematologic (absolute neutrophil count ≥ 1.5x109/L, hemoglobin concentration ≥ 90g/L, platelet count ≥ 100 x109/L), hepatic (albumin ≥ 28 g/L, total bilirubin < 1.5 times the upper limit of normal (ULN), alanine aminotransferase and aspartate aminotransferase < 5×ULN) and renal function (serum creatine < 1.5×ULN, creatinine clearance rate ≥ 45ml/min);
8. Life expectancy of at least 12 weeks.

Exclusion Criteria:

1. Have acute or chronic active hepatitis B or C, HBV-DNA>2000IU/ml or 104 copy/ml; HCV-RNA>103 copy/ml; both HBsAg and HCV antibody are positive. If the related results become lower than above standards after anti-viral treatment, the patients are qualified for enrolment;
2. Have metastasis in extrahepatic distant organs including lung, central nervous system, bone and etc. Or extrahepatic lymph node metastasis beyond abdomen;
3. Have risky bleeding events requiring transfusion, operation or local therapies, continuous medication in the past 3 months;
4. Have thromboembolism in the past 6 months, including myocardial infarction, unstable angina, stroke or transient ischemic attack, pulmonary embolism, deep vein thrombosis;
5. Have taken aspirin (>325mg/day) or other antiplatelet drugs continuously for 10 days or more within 2 weeks before enrolment;
6. Uncontrollable hypertension, systolic pressure>140mmHg or diastolic pressure>90mmHg after best medical care, or history of hypertensive crisis or hypertensive encephalopathy;
7. Symptomatic congestive heart failure (NYHA class II-IV). Symptomatic or badly-controlled arrhythmia. Congenital long QT syndrome or modified QTc>500ms upon screening;
8. Have active autoimmune diseases that require systemic treatment within 2 years before enrolment;
9. Active tuberculosis, having antituberculosis therapy at present or within 1 year;
10. Have a known history of prior invasive malignancies within 5 years before enrolment;
11. Pregnant or breastfeeding women, or expecting to conceive or father children within the projected duration of the trial;
12. Have other uncontrollable comorbidities;
13. Infection of HIV, known syphilis requiring treatment;
14. Allergic to elements of camrelizumab.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival, PFS | one years
  defined as the time from the commencement of radiotherapy until disease progression or death from any cause, whichever happens first. Patients who withdraw or who are lost to follow-up will be censored at the date of the last adequate tumor assessment. Patients not having an event will be censored at the date of the last adequate tumor assessment. If patients don't have baseline tumor assessments, they will be censored at the date of the first treatment.

SECONDARY OUTCOMES:
Overall survival, OS | one years
  defined as the time from the commencement of radiotherapy until death from any cause. Patients who withdraw or are lost to follow-up or still alive will be at the date last known to be alive.
Adverse events, AE | one years
  adverse events during the treatment period using Common Terminology Criteria for Adverse Events (CTCAE) (version 5.0).
Objective response rate, ORR | one years
  defined as the proportion of participants with a complete response or partial response according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.1.
Disease control rate, DCR | one years
  defined as the proportion of participants with a complete response, partial response, or stable disease according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Kuang, PhD, Study Chair — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhu M, Jin M, Zhao X, Shen S, Chen Y, Xiao H, Wei G, He Q, Li B, Peng Z. Anti-PD-1 antibody in combination with radiotherapy as first-line therapy for unresectable intrahepatic cholangiocarcinoma. BMC Med. 2024 Apr 19;22(1):165. doi: 10.1186/s12916-024-03381-4. PMID 38637772